CLINICAL TRIAL: NCT02716675
Title: A Phase 2b Study to Evaluate the Safety and Efficacy of VRC01 Broadly Neutralizing Monoclonal Antibody in Reducing Acquisition of HIV-1 Infection Among Men and Transgender Persons Who Have Sex With Men
Brief Title: Evaluating the Safety and Efficacy of the VRC01 Antibody in Reducing Acquisition of HIV-1 Infection Among Men and Transgender Persons Who Have Sex With Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 704/HPTN 085; 30095 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: HIV Infections
Keywords: HIV-1 Infections
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Low-Dose VRC01 (Experimental): Participants will receive an intravenous (IV) infusion of 10 mg/kg of VRC01 over about 15 to 60 minutes at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.
  Interventions: Biological: VRC01
- Group 2: High-Dose VRC01 (Experimental): Participants will receive an IV infusion of 30 mg/kg of VRC01 over about 15 to 60 minutes at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.
  Interventions: Biological: VRC01
- Group 3: VRC01 Placebo (Placebo Comparator): Participants will receive an IV infusion of placebo for VRC01 over about 15 to 60 minutes at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.
  Interventions: Biological: Placebo for VRC01

INTERVENTIONS:
Biological: VRC01 — Administered by IV infusion; total dose will vary based on participant's weight
  Other Names: Human monoclonal antibody (mAb) VRC-HIVMAB060-00-AB
  Arms: Group 1: Low-Dose VRC01; Group 2: High-Dose VRC01
Biological: Placebo for VRC01 — Sodium Chloride for Injection USP, 0.9%; administered by IV infusion
  Arms: Group 3: VRC01 Placebo

SUMMARY:
This study will evaluate the safety and efficacy of the human monoclonal antibody (mAb) VRC-HIVMAB060-00-AB (VRC01) in preventing HIV-1 infection among men and transgender (TG) persons who have sex with men, in North America, South America, and Switzerland.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and efficacy of the VRC01 antibody in preventing HIV-1 infection in men and transgender (TG) persons who have sex with men, in North America, South America, and Switzerland.

Participants will be randomized to receive VRC01 mAb by intravenous (IV) infusion at a dose of 10 mg/kg or 30 mg/kg every 8 weeks, or to receive control infusions every 8 weeks. All participants will receive the VRC01 antibody or placebo by IV infusion at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72. For 3 days following each infusion, participants will be asked to record and report any symptoms to study researchers.

In addition to the infusion visits, participants will attend study visits at Weeks 4, 8 + 5 days, 12, 20, 28, 36, 44, 52, 60, 68, 76, 80, 88, 96, and 104. All study visits will include blood collection and HIV testing and counseling. Select study visits will include a medical history review, physical exam, urine collection, pregnancy testing for participants capable of becoming pregnant, risk reduction counseling, and an interview/questionnaire.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study and completes a questionnaire prior to first infusion with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent for the duration of the participant's trial participation
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Persons born Male or identifying as Transgender (TG) (male-to-female or female-to-male, see HVTN 704/HPTN 085 SSP) who, in the 6 months prior to randomization, experienced 1 or both of the following HIV risk criteria:

  * Condomless anal intercourse with 1 or more male or transgender partner(s)
  * Anal intercourse with 2 or more male or transgender partners
* Male-to-female and female-to-male TG volunteers are eligible. Receipt of hormonal therapy does not make a TG volunteer ineligible.
* Volunteers who have been in a mutually monogamous relationship with an HIV-1 seronegative partner for greater than 1 year are excluded.

Laboratory Inclusion Values:

Hematology

* Hemoglobin (Hgb) greater than or equal to 10.5 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male (greater than or equal to 12.0 g/dL for transgender women taking feminizing hormones [e.g., anti-androgens, estrogens])
* Platelets greater than or equal to 100,000 cells/mm^3

Chemistry

* Alanine aminotransferase (ALT) less than 2.5 times the institutional upper limit of normal and creatinine less than or equal to 1.25 times the institutional upper limit of normal

Virology

* HIV uninfected, as defined in the SSP, within 30 days prior to enrollment

Urine

* Negative, trace, or 1+ (30 g/L for semi-quantitative) urine protein by dipstick

Reproductive Status

* Volunteers capable of becoming pregnant: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed at the screening visit and prior to infusion on the day of initial infusion. Persons who are NOT capable of becoming pregnant due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records) are not required to undergo pregnancy testing.
* Reproductive Status: A volunteer who is capable of becoming pregnant must agree to consistently use effective contraception (see the protocol and SSP for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit.
* Volunteers capable of becoming pregnant must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Investigational research agents received within 30 days before first infusion
* Body mass index (BMI) greater than or equal to 40
* Pregnant or breastfeeding
* Any reactive, indeterminate, or positive HIV test, even if subsequent testing indicates that the individual is not HIV infected, except as permitted by the HVTN 704/HPTN 085 Protocol Safety Review Team (PSRT).

Vaccines

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 704/HPTN 085 PSRT will determine eligibility on a case-by-case basis.

Immune System

* Serious adverse reactions to VRC01 formulation components such as sodium citrate, sodium chloride, and L-arginine hydrochloride, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
* Autoimmune disease, including Type I diabetes mellitus (Not excluded from participation: Volunteer with mild, stable and uncomplicated autoimmune disease that does not require consistent immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate reactogenicity and AE assessments)
* Immunodeficiency syndrome

Clinically Significant Medical Conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * Any contraindication to repeated infusions or blood draws, including inability to establish venous access;
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period; or
  * A condition or process for which signs or symptoms could be confused with reactions to VRC01.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or infusion reactions, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Asthma, other than mild, well-controlled asthma
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* History of receiving transplantation of life-saving organs or tissues (includes heart, kidney, pancreas, lungs, liver, and intestines)
* Known hepatic or renal dysfunction

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2699 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Corey, Study Chair — HVTN; FHCRC; Myron Cohen, Study Chair — HPTN; University of North Carolina
Locations (26):
- United States (19):
  - Alabama CRS, Birmingham, Alabama
  - UCLA Vine Street Clinic CRS, Los Angeles, California
  - Bridge HIV CRS, San Francisco, California
  - George Washington Univ. CRS, Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Harlem Prevention Center CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Bronx Prevention Research Center CRS, The Bronx, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Peru (5):
  - ACSA CRS, Iquitos, Maynas
  - CITBM - UNIDEC, Centro de Investigaciones Tecnológicas, Biomédicas y Medioambientales CRS, Bellavista, Provincia Constitucional del Callao
  - Barranco CRS, Lima
  - San Miguel CRS, Lima
  - Via Libre CRS, Lima
- Lausanne Vaccine and Immunotherapy Center CRS, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Edupuganti S, Mgodi N, Karuna ST, Andrew P, Rudnicki E, Kochar N, deCamp A, De La Grecca R, Anderson M, Karg C, Tindale I, Greene E, Broder GB, Lucas J, Hural J, Gallardo-Cartagena JA, Gonzales P, Frank I, Sobieszczyk M, Gomez Lorenzo MM, Burns D, Anderson PL, Miner MD, Ledgerwood J, Mascola JR, Gilbert PB, Cohen MS, Corey L; HVTN 704/HPTN 085 study group. Feasibility and Successful Enrollment in a Proof-of-Concept HIV Prevention Trial of VRC01, a Broadly Neutralizing HIV-1 Monoclonal Antibody. J Acquir Immune Defic Syndr. 2021 May 1;87(1):671-679. doi: 10.1097/QAI.0000000000002639. PMID 33587505
- [Result] Mgodi NM, Takuva S, Edupuganti S, Karuna S, Andrew P, Lazarus E, Garnett P, Shava E, Mukwekwerere PG, Kochar N, Marshall K, Rudnicki E, Juraska M, Anderson M, Karg C, Tindale I, Greene E, Luthuli N, Baepanye K, Hural J, Gomez Lorenzo MM, Burns D, Miner MD, Ledgerwood J, Mascola JR, Donnell D, Cohen MS, Corey L; HVTN 703/HPTN 081 Team. A Phase 2b Study to Evaluate the Safety and Efficacy of VRC01 Broadly Neutralizing Monoclonal Antibody in Reducing Acquisition of HIV-1 Infection in Women in Sub-Saharan Africa: Baseline Findings. J Acquir Immune Defic Syndr. 2021 May 1;87(1):680-687. doi: 10.1097/QAI.0000000000002649. PMID 33587510
- [Result] Huang Y, Naidoo L, Zhang L, Carpp LN, Rudnicki E, Randhawa A, Gonzales P, McDermott A, Ledgerwood J, Lorenzo MMG, Burns D, DeCamp A, Juraska M, Mascola J, Edupuganti S, Mgodi N, Cohen M, Corey L, Andrew P, Karuna S, Gilbert PB, Mngadi K, Lazarus E. Pharmacokinetics and predicted neutralisation coverage of VRC01 in HIV-uninfected participants of the Antibody Mediated Prevention (AMP) trials. EBioMedicine. 2021 Feb;64:103203. doi: 10.1016/j.ebiom.2020.103203. Epub 2021 Jan 23. PMID 33493795
- [Result] Huang Y, Zhang L, Eaton A, Mkhize NN, Carpp LN, Rudnicki E, DeCamp A, Juraska M, Randhawa A, McDermott A, Ledgerwood J, Andrew P, Karuna S, Edupuganti S, Mgodi N, Cohen M, Corey L, Mascola J, Gilbert PB, Morris L, Montefiori DC. Prediction of serum HIV-1 neutralization titers of VRC01 in HIV-uninfected Antibody Mediated Prevention (AMP) trial participants. Hum Vaccin Immunother. 2022 Dec 31;18(1):1908030. doi: 10.1080/21645515.2021.1908030. Epub 2021 Jul 2. PMID 34213402
- [Result] Corey L, Gilbert PB, Juraska M, Montefiori DC, Morris L, Karuna ST, Edupuganti S, Mgodi NM, deCamp AC, Rudnicki E, Huang Y, Gonzales P, Cabello R, Orrell C, Lama JR, Laher F, Lazarus EM, Sanchez J, Frank I, Hinojosa J, Sobieszczyk ME, Marshall KE, Mukwekwerere PG, Makhema J, Baden LR, Mullins JI, Williamson C, Hural J, McElrath MJ, Bentley C, Takuva S, Gomez Lorenzo MM, Burns DN, Espy N, Randhawa AK, Kochar N, Piwowar-Manning E, Donnell DJ, Sista N, Andrew P, Kublin JG, Gray G, Ledgerwood JE, Mascola JR, Cohen MS; HVTN 704/HPTN 085 and HVTN 703/HPTN 081 Study Teams. Two Randomized Trials of Neutralizing Antibodies to Prevent HIV-1 Acquisition. N Engl J Med. 2021 Mar 18;384(11):1003-1014. doi: 10.1056/NEJMoa2031738. PMID 33730454
- [Derived] Reeves DB, Mayer BT, deCamp AC, Huang Y, Zhang B, Carpp LN, Magaret CA, Juraska M, Gilbert PB, Montefiori DC, Bar KJ, Cardozo-Ojeda EF, Schiffer JT, Rossenkhan R, Edlefsen P, Morris L, Mkhize NN, Williamson C, Mullins JI, Seaton KE, Tomaras GD, Andrew P, Mgodi N, Ledgerwood JE, Cohen MS, Corey L, Naidoo L, Orrell C, Goepfert PA, Casapia M, Sobieszczyk ME, Karuna ST, Edupuganti S. High monoclonal neutralization titers reduced breakthrough HIV-1 viral loads in the Antibody Mediated Prevention trials. Nat Commun. 2023 Dec 14;14(1):8299. doi: 10.1038/s41467-023-43384-y. PMID 38097552
- [Derived] Huang Y, Zhang L, Karuna S, Andrew P, Juraska M, Weiner JA, Angier H, Morgan E, Azzam Y, Swann E, Edupuganti S, Mgodi NM, Ackerman ME, Donnell D, Gama L, Anderson PL, Koup RA, Hural J, Cohen MS, Corey L, McElrath MJ, Gilbert PB, Lemos MP. Adults on pre-exposure prophylaxis (tenofovir-emtricitabine) have faster clearance of anti-HIV monoclonal antibody VRC01. Nat Commun. 2023 Nov 28;14(1):7813. doi: 10.1038/s41467-023-43399-5. PMID 38016958

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned to the placebo, low-dose VRC01, or high-dose VRC01 arm. The pooled VRC01 arm represents participants assigned to low-dose or high-dose VRC01 and is the primary comparison group for the primary analysis of prevention efficacy.
Groups:
- Placebo: Placebo (Sodium Chloride, USP 0.9%) by intravenous (IV) infusion at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
- Low-Dose VRC01: VRC01 mAb by intravenous (IV) infusion at a dose of 10 mg/kg at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
- High-Dose VRC01: VRC01 mAb by intravenous (IV) infusion at a dose of 30 mg/kg at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
Period: Overall Study
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01
Started (Enrollment is concurrent with receiving the first infusion (safety analyses)) | 903 | 899 | 897
Modified Intent-to-treat Population (Participants excluded from MITT if HIV positive at enrollment or randomized/enrolled more than once (efficacy analyses)) | 898 | 895 | 894
Completed | 703 | 702 | 686
Not Completed | 200 | 197 | 211
Not completed — Death | 2 | 3 | 0
Not completed — Physician Decision | 2 | 1 | 1
Not completed — Lost to Follow-up | 100 | 87 | 99
Not completed — Withdrawal by Subject | 22 | 25 | 20
Not completed — Protocol Violation | 0 | 3 | 1
Not completed — Participant Unable to Adhere to Visit Schedule | 36 | 31 | 42
Not completed — Other | 38 | 47 | 48

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Total
Number analyzed (Participants) | 903 | 899 | 897 | 2699
Age, Continuous [Median (Full Range); unit: years] | 28 [18 to 50] | 28 [18 to 52] | 27 [18 to 50] | 28 [18 to 52]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0
  18 - 20 years | 95 | 94 | 106 | 295
  21 - 30 years | 496 | 474 | 480 | 1450
  31 - 40 years | 232 | 253 | 208 | 693
  41 - 50 years | 80 | 77 | 103 | 260
  Above 50 years | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 8 | 26
  Male | 892 | 892 | 889 | 2673
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 532 | 517 | 495 | 1544
  Not Hispanic or Latino | 371 | 382 | 402 | 1155
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 7 | 3 | 16
  Asian | 22 | 29 | 18 | 69
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 2 | 8
  Black or African American | 132 | 132 | 144 | 408
  White | 286 | 272 | 293 | 851
  More than one race | 32 | 32 | 24 | 88
  Unknown or Not Reported | 421 | 425 | 413 | 1259
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 460 | 464 | 457 | 1381
  Brazil | 51 | 49 | 51 | 151
  Peru | 380 | 374 | 377 | 1131
  Switzerland | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured through 3 days after each infusion at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Pooled VRC01: VRC01 mAb by intravenous (IV) infusion at a dose of 10 or 30 mg/kg at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
Participants
  Pain: None | 812 | 794 | 805 | 1599
  Pain: Mild | 90 | 104 | 88 | 192
  Pain: Moderate | 1 | 1 | 4 | 5
  Pain: Severe | 0 | 0 | 0 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0
  Tenderness: None | 754 | 741 | 759 | 1500
  Tenderness: Mild | 145 | 153 | 133 | 286
  Tenderness: Moderate | 4 | 5 | 5 | 10
  Tenderness: Severe | 0 | 0 | 0 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 718 | 702 | 720 | 1422
  Pain and/or Tenderness: Mild | 180 | 191 | 170 | 361
  Pain and/or Tenderness: Moderate | 5 | 6 | 7 | 13
  Pain and/or Tenderness: Severe | 0 | 0 | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 3 days after each infusion at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
Participants
  Erythema/Redness: None | 877 | 878 | 882 | 1760
  Erythema/Redness: Gr 1: 2.5 to less than 5cm | 17 | 13 | 13 | 26
  Erythema/Redness: Gr 2: 5 to less than 10cm | 9 | 8 | 2 | 10
  Erythema/Redness: Gr 3: >= 10cm | 0 | 0 | 0 | 0
  Erythema/Redness: Gr 4: complications AE | 0 | 0 | 0 | 0
  Erythema/Redness: Missing | 0 | 0 | 0 | 0
  Induration/Swelling: None | 896 | 894 | 894 | 1788
  Induration/Swelling: Gr 1: 2.5 to less than 5cm | 7 | 4 | 2 | 6
  Induration/Swelling: Gr 2: 5 to less than 10cm | 0 | 1 | 1 | 2
  Induration/Swelling: Gr 3: >= 10cm | 0 | 0 | 0 | 0
  Induration/Swelling: Gr 4: complications AE | 0 | 0 | 0 | 0
  Induration/Swelling: Missing | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 874 | 876 | 880 | 1756
  Erythema and/or Induration: Gr 1: 2.5 to less than 5cm | 20 | 15 | 14 | 29
  Erythema and/or Induration: Gr 2: 5 to less than 10cm | 9 | 8 | 3 | 11
  Erythema and/or Induration: Gr 3: >= 10cm | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 4: complications AE | 0 | 0 | 0 | 0
  Erythema and/or Induration: Missing | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Symptoms is the maximum of the individual systemic reactogenicities excluding body temperature for a participant.
Time Frame: Measured through 3 days after each infusion at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
Participants
  Malaise and/or fatigue: None | 664 | 672 | 691 | 1363
  Malaise and/or fatigue: Mild | 197 | 182 | 169 | 351
  Malaise and/or fatigue: Moderate | 39 | 45 | 36 | 81
  Malaise and/or fatigue: Severe | 3 | 0 | 1 | 1
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 809 | 802 | 820 | 1622
  Myalgia: Mild | 81 | 76 | 61 | 137
  Myalgia: Moderate | 13 | 21 | 15 | 36
  Myalgia: Severe | 0 | 0 | 1 | 1
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Headache: None | 728 | 714 | 731 | 1445
  Headache: Mild | 146 | 147 | 137 | 284
  Headache: Moderate | 28 | 35 | 29 | 64
  Headache: Severe | 1 | 3 | 0 | 3
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 821 | 814 | 812 | 1626
  Nausea: Mild | 74 | 74 | 77 | 151
  Nausea: Moderate | 8 | 10 | 8 | 18
  Nausea: Severe | 0 | 1 | 0 | 1
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0
  Vomiting: None | 889 | 873 | 881 | 1754
  Vomiting: Mild | 12 | 24 | 12 | 36
  Vomiting: Moderate | 2 | 2 | 4 | 6
  Vomiting: Severe | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0
  Chills: None | 857 | 843 | 861 | 1704
  Chills: Mild | 41 | 45 | 29 | 74
  Chills: Moderate | 5 | 11 | 6 | 17
  Chills: Severe | 0 | 0 | 1 | 1
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0
  Arthralgia: None | 861 | 848 | 869 | 1717
  Arthralgia: Mild | 39 | 44 | 21 | 65
  Arthralgia: Moderate | 3 | 7 | 7 | 14
  Arthralgia: Severe | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 556 | 546 | 563 | 1109
  Max. Systemic Symptoms: Mild | 286 | 277 | 273 | 550
  Max. Systemic Symptoms: Moderate | 57 | 72 | 59 | 131
  Max. Systemic Symptoms: Severe | 4 | 4 | 2 | 6
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0
  Increased Body Temperature: None | 880 | 879 | 870 | 1749
  Increased Body Temperature: Mild | 14 | 11 | 14 | 25
  Increased Body Temperature: Moderate | 7 | 7 | 12 | 19
  Increased Body Temperature: Severe | 1 | 2 | 1 | 3
  Increased Body Temperature: Potentially Life-threatening | 1 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alanine Aminotransferase (ALT)
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: Safety population. Participants may not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
U/L
  ALT (SGPT) (U/L)- Week 0 | 25 [17 to 35] | 24 [17 to 36] | 24 [17 to 35] | 24 [17 to 35]
  ALT (SGPT) (U/L)- Week 8: number analyzed (Participants) | 865 | 855 | 856 | 1711
  ALT (SGPT) (U/L)- Week 8 | 24 [17 to 35] | 24 [16 to 36] | 24 [17 to 33] | 24 [17 to 35]
  ALT (SGPT) (U/L)- Week 16: number analyzed (Participants) | 841 | 836 | 832 | 1668
  ALT (SGPT) (U/L)- Week 16 | 23 [17 to 35] | 23 [17 to 34] | 24 [17 to 34] | 23 [17 to 34]
  ALT (SGPT) (U/L)- Week 24: number analyzed (Participants) | 811 | 820 | 805 | 1625
  ALT (SGPT) (U/L)- Week 24 | 24 [17 to 35] | 23 [17 to 33] | 23 [16 to 33] | 23 [16 to 33]
  ALT (SGPT) (U/L)- Week 32: number analyzed (Participants) | 802 | 797 | 787 | 1584
  ALT (SGPT) (U/L)- Week 32 | 24 [17 to 34] | 23 [17 to 34] | 23 [16 to 33] | 23 [16 to 33]
  ALT (SGPT) (U/L)- Week 40: number analyzed (Participants) | 790 | 784 | 765 | 1549
  ALT (SGPT) (U/L)- Week 40 | 23 [16 to 33] | 22 [16 to 33] | 22 [16 to 33] | 22 [16 to 33]
  ALT (SGPT) (U/L)- Week 48: number analyzed (Participants) | 772 | 776 | 754 | 1530
  ALT (SGPT) (U/L)- Week 48 | 23 [16 to 33] | 23 [16 to 33] | 22 [15 to 31] | 22 [16 to 32]
  ALT (SGPT) (U/L)- Week 56: number analyzed (Participants) | 754 | 763 | 749 | 1512
  ALT (SGPT) (U/L)- Week 56 | 22 [16 to 34] | 22 [16 to 33] | 22 [16 to 30] | 22 [16 to 32]
  ALT (SGPT) (U/L)- Week 64: number analyzed (Participants) | 737 | 748 | 722 | 1470
  ALT (SGPT) (U/L)- Week 64 | 22 [16 to 33] | 22 [16 to 33] | 22 [15 to 31] | 22 [16 to 32]
  ALT (SGPT) (U/L)- Week 72: number analyzed (Participants) | 721 | 731 | 718 | 1449
  ALT (SGPT) (U/L)- Week 72 | 22 [16 to 32] | 22 [16 to 31] | 22 [16 to 31] | 22 [16 to 31]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
mg/dL
  Creatinine (mg/dL)- Week 0 | 0.86 [0.76 to 0.98] | 0.86 [0.75 to 0.97] | 0.86 [0.76 to 0.99] | 0.86 [0.75 to 0.98]
  Creatinine (mg/dL)- Week 8: number analyzed (Participants) | 866 | 855 | 856 | 1711
  Creatinine (mg/dL)- Week 8 | 0.87 [0.77 to 0.98] | 0.86 [0.76 to 0.97] | 0.88 [0.77 to 0.99] | 0.87 [0.77 to 0.98]
  Creatinine (mg/dL)- Week 16: number analyzed (Participants) | 841 | 836 | 832 | 1668
  Creatinine (mg/dL)- Week 16 | 0.88 [0.78 to 0.99] | 0.87 [0.77 to 0.98] | 0.87 [0.78 to 0.99] | 0.87 [0.77 to 0.99]
  Creatinine (mg/dL)- Week 24: number analyzed (Participants) | 812 | 820 | 805 | 1625
  Creatinine (mg/dL)- Week 24 | 0.87 [0.77 to 0.99] | 0.88 [0.78 to 0.99] | 0.88 [0.77 to 1] | 0.88 [0.77 to 1]
  Creatinine (mg/dL)- Week 32: number analyzed (Participants) | 802 | 797 | 787 | 1584
  Creatinine (mg/dL)- Week 32 | 0.88 [0.77 to 0.99] | 0.87 [0.78 to 0.99] | 0.87 [0.77 to 1] | 0.87 [0.78 to 0.99]
  Creatinine (mg/dL)- Week 40: number analyzed (Participants) | 791 | 786 | 765 | 1551
  Creatinine (mg/dL)- Week 40 | 0.88 [0.78 to 0.99] | 0.88 [0.78 to 1] | 0.88 [0.78 to 1] | 0.88 [0.78 to 1]
  Creatinine (mg/dL)- Week 48: number analyzed (Participants) | 772 | 776 | 754 | 1530
  Creatinine (mg/dL)- Week 48 | 0.88 [0.78 to 1] | 0.89 [0.79 to 0.99] | 0.89 [0.78 to 1.01] | 0.89 [0.79 to 1]
  Creatinine (mg/dL)- Week 56: number analyzed (Participants) | 754 | 763 | 750 | 1513
  Creatinine (mg/dL)- Week 56 | 0.88 [0.78 to 0.99] | 0.89 [0.78 to 1] | 0.88 [0.8 to 1] | 0.88 [0.79 to 1]
  Creatinine (mg/dL)- Week 64: number analyzed (Participants) | 737 | 748 | 722 | 1470
  Creatinine (mg/dL)- Week 64 | 0.88 [0.78 to 1] | 0.89 [0.8 to 1] | 0.89 [0.79 to 1] | 0.89 [0.79 to 1]
  Creatinine (mg/dL)- Week 72: number analyzed (Participants) | 722 | 732 | 718 | 1450
  Creatinine (mg/dL)- Week 72 | 0.89 [0.79 to 0.99] | 0.88 [0.8 to 1] | 0.89 [0.8 to 1.01] | 0.89 [0.8 to 1]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
g/dL
  Hemoglobin (g/dL)- Week 0: number analyzed (Participants) | 902 | 899 | 897 | 1796
  Hemoglobin (g/dL)- Week 0 | 14.9 [14.1 to 15.6] | 14.8 [14.2 to 15.6] | 14.9 [14.1 to 15.6] | 14.8 [14.2 to 15.6]
  Hemoglobin (g/dL)- Week 8: number analyzed (Participants) | 865 | 853 | 855 | 1708
  Hemoglobin (g/dL)- Week 8 | 14.7 [14.1 to 15.5] | 14.7 [13.9 to 15.4] | 14.8 [14.1 to 15.5] | 14.7 [14 to 15.4]
  Hemoglobin (g/dL)- Week 16: number analyzed (Participants) | 841 | 836 | 832 | 1668
  Hemoglobin (g/dL)- Week 16 | 14.7 [14 to 15.5] | 14.7 [14 to 15.4] | 14.7 [14 to 15.4] | 14.7 [14 to 15.4]
  Hemoglobin (g/dL)- Week 24: number analyzed (Participants) | 812 | 819 | 805 | 1624
  Hemoglobin (g/dL)- Week 24 | 14.6 [14 to 15.4] | 14.6 [13.9 to 15.3] | 14.7 [14 to 15.3] | 14.7 [14 to 15.3]
  Hemoglobin (g/dL)- Week 32: number analyzed (Participants) | 802 | 797 | 788 | 1585
  Hemoglobin (g/dL)- Week 32 | 14.6 [14 to 15.3] | 14.6 [13.9 to 15.3] | 14.7 [13.9 to 15.3] | 14.6 [13.9 to 15.3]
  Hemoglobin (g/dL)- Week 40: number analyzed (Participants) | 790 | 786 | 765 | 1551
  Hemoglobin (g/dL)- Week 40 | 14.6 [13.9 to 15.5] | 14.5 [13.8 to 15.3] | 14.6 [13.9 to 15.4] | 14.6 [13.8 to 15.3]
  Hemoglobin (g/dL)- Week 48: number analyzed (Participants) | 772 | 775 | 753 | 1528
  Hemoglobin (g/dL)- Week 48 | 14.6 [13.9 to 15.4] | 14.6 [13.8 to 15.3] | 14.6 [13.8 to 15.3] | 14.6 [13.8 to 15.3]
  Hemoglobin (g/dL)- Week 56: number analyzed (Participants) | 754 | 763 | 750 | 1513
  Hemoglobin (g/dL)- Week 56 | 14.6 [13.9 to 15.4] | 14.6 [13.7 to 15.3] | 14.6 [13.9 to 15.3] | 14.6 [13.8 to 15.3]
  Hemoglobin (g/dL)- Week 64: number analyzed (Participants) | 737 | 748 | 721 | 1469
  Hemoglobin (g/dL)- Week 64 | 14.6 [13.8 to 15.3] | 14.5 [13.7 to 15.4] | 14.6 [13.8 to 15.3] | 14.5 [13.8 to 15.3]
  Hemoglobin (g/dL)- Week 72: number analyzed (Participants) | 722 | 731 | 719 | 1450
  Hemoglobin (g/dL)- Week 72 | 14.5 [13.9 to 15.3] | 14.5 [13.7 to 15.2] | 14.5 [13.8 to 15.3] | 14.5 [13.7 to 15.3]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: cells/cubic mm
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
cells/cubic mm
  Lymphocytes (cells/cubic mm)- Week 0: number analyzed (Participants) | 902 | 899 | 897 | 1796
  Lymphocytes (cells/cubic mm)- Week 0 | 1988.5 [1620 to 2363] | 1980 [1600 to 2406] | 1971 [1645 to 2370] | 1978.5 [1620 to 2392]
  Lymphocytes (cells/cubic mm)- Week 8: number analyzed (Participants) | 865 | 851 | 854 | 1705
  Lymphocytes (cells/cubic mm)- Week 8 | 1926 [1610 to 2296] | 1904 [1571 to 2264] | 1947.5 [1596 to 2310] | 1930 [1590 to 2294]
  Lymphocytes (cells/cubic mm)- Week 16: number analyzed (Participants) | 840 | 836 | 832 | 1668
  Lymphocytes (cells/cubic mm)- Week 16 | 1927.5 [1600 to 2289] | 1896 [1593.5 to 2325.5] | 1915.5 [1592 to 2349.5] | 1900.5 [1593 to 2339]
  Lymphocytes (cells/cubic mm)- Week 24: number analyzed (Participants) | 811 | 819 | 805 | 1624
  Lymphocytes (cells/cubic mm)- Week 24 | 1950 [1600 to 2295] | 1925 [1580 to 2320] | 1911 [1600 to 2336] | 1920 [1596 to 2330.5]
  Lymphocytes (cells/cubic mm)- Week 32: number analyzed (Participants) | 802 | 797 | 788 | 1585
  Lymphocytes (cells/cubic mm)- Week 32 | 1957 [1610 to 2300] | 1930 [1560 to 2300] | 1900 [1580 to 2309.5] | 1920 [1570 to 2304]
  Lymphocytes (cells/cubic mm)- Week 40: number analyzed (Participants) | 789 | 786 | 765 | 1551
  Lymphocytes (cells/cubic mm)- Week 40 | 1890 [1560 to 2294] | 1900 [1525 to 2295] | 1879 [1570 to 2250] | 1890 [1550 to 2263]
  Lymphocytes (cells/cubic mm)- Week 48: number analyzed (Participants) | 772 | 774 | 752 | 1526
  Lymphocytes (cells/cubic mm)- Week 48 | 1923.5 [1600 to 2271] | 1923 [1570 to 2320] | 1870 [1570 to 2260] | 1900 [1570 to 2290]
  Lymphocytes (cells/cubic mm)- Week 56: number analyzed (Participants) | 754 | 762 | 750 | 1512
  Lymphocytes (cells/cubic mm)- Week 56 | 1910 [1582 to 2290] | 1887.5 [1565 to 2310] | 1900.5 [1600 to 2294] | 1895.5 [1582.5 to 2300]
  Lymphocytes (cells/cubic mm)- Week 64: number analyzed (Participants) | 737 | 748 | 721 | 1469
  Lymphocytes (cells/cubic mm)- Week 64 | 1922 [1593 to 2300] | 1890 [1580 to 2311] | 1870 [1570 to 2260] | 1880 [1580 to 2300]
  Lymphocytes (cells/cubic mm)- Week 72: number analyzed (Participants) | 722 | 731 | 719 | 1450
  Lymphocytes (cells/cubic mm)- Week 72 | 1940 [1590 to 2236] | 1930 [1542 to 2267] | 1900 [1560 to 2280] | 1910 [1556 to 2270]
  Neutrophils (cells/cubic mm)- Week 0: number analyzed (Participants) | 902 | 899 | 897 | 1796
  Neutrophils (cells/cubic mm)- Week 0 | 3586 [2754 to 4495] | 3593 [2720 to 4514] | 3534 [2705 to 4505] | 3571.5 [2715 to 4510.5]
  Neutrophils (cells/cubic mm)- Week 8: number analyzed (Participants) | 865 | 851 | 854 | 1705
  Neutrophils (cells/cubic mm)- Week 8 | 3410 [2727 to 4236] | 3460 [2650 to 4540] | 3424 [2798 to 4460] | 3437 [2708 to 4502]
  Neutrophils (cells/cubic mm)- Week 16: number analyzed (Participants) | 840 | 836 | 832 | 1668
  Neutrophils (cells/cubic mm)- Week 16 | 3378 [2578 to 4355] | 3377 [2549.5 to 4246] | 3360 [2600 to 4305] | 3361.5 [2580 to 4283]
  Neutrophils (cells/cubic mm)- Week 24: number analyzed (Participants) | 811 | 819 | 805 | 1624
  Neutrophils (cells/cubic mm)- Week 24 | 3330 [2610 to 4212] | 3417 [2554 to 4430] | 3306 [2538 to 4350] | 3357.5 [2550 to 4400]
  Neutrophils (cells/cubic mm)- Week 32: number analyzed (Participants) | 802 | 797 | 788 | 1585
  Neutrophils (cells/cubic mm)- Week 32 | 3344 [2543 to 4300] | 3360 [2501 to 4380] | 3336 [2582.5 to 4289] | 3350 [2550 to 4352]
  Neutrophils (cells/cubic mm)- Week 40: number analyzed (Participants) | 789 | 786 | 765 | 1551
  Neutrophils (cells/cubic mm)- Week 40 | 3310 [2560 to 4195] | 3260 [2500 to 4400] | 3300 [2516 to 4200] | 3287 [2500 to 4320]
  Neutrophils (cells/cubic mm)- Week 48: number analyzed (Participants) | 772 | 774 | 752 | 1526
  Neutrophils (cells/cubic mm)- Week 48 | 3322 [2675 to 4344.5] | 3284.5 [2560 to 4240] | 3266.5 [2583 to 4205] | 3278 [2580 to 4224]
  Neutrophils (cells/cubic mm)- Week 56: number analyzed (Participants) | 754 | 762 | 750 | 1512
  Neutrophils (cells/cubic mm)- Week 56 | 3340 [2612 to 4320] | 3238.5 [2500 to 4290] | 3200 [2519 to 4100] | 3212.5 [2508 to 4192.5]
  Neutrophils (cells/cubic mm)- Week 64: number analyzed (Participants) | 737 | 748 | 721 | 1469
  Neutrophils (cells/cubic mm)- Week 64 | 3245 [2560 to 4180] | 3240 [2495 to 4275] | 3228 [2576 to 4100] | 3230 [2520 to 4190]
  Neutrophils (cells/cubic mm)- Week 72: number analyzed (Participants) | 722 | 731 | 719 | 1450
  Neutrophils (cells/cubic mm)- Week 72 | 3286.5 [2530 to 4123] | 3245 [2420 to 4180] | 3304 [2550 to 4298] | 3272 [2500 to 4259]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, White Blood Cells (WBC)
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
1000 cells/cubic mm
  WBC (1000 cells/cubic mm)- Week 0: number analyzed (Participants) | 902 | 899 | 897 | 1796
  WBC (1000 cells/cubic mm)- Week 0 | 6.33 [5.28 to 7.5] | 6.4 [5.28 to 7.66] | 6.3 [5.2 to 7.5] | 6.3 [5.25 to 7.6]
  WBC (1000 cells/cubic mm)- Week 8: number analyzed (Participants) | 865 | 853 | 855 | 1708
  WBC (1000 cells/cubic mm)- Week 8 | 6.2 [5.2 to 7.4] | 6.1 [5.01 to 7.41] | 6.2 [5.1 to 7.5] | 6.12 [5.07 to 7.5]
  WBC (1000 cells/cubic mm)- Week 16: number analyzed (Participants) | 841 | 836 | 832 | 1668
  WBC (1000 cells/cubic mm)- Week 16 | 6.1 [4.99 to 7.3] | 6.1 [5 to 7.3] | 6.1 [5.01 to 7.33] | 6.1 [5 to 7.3]
  WBC (1000 cells/cubic mm)- Week 24: number analyzed (Participants) | 812 | 819 | 805 | 1624
  WBC (1000 cells/cubic mm)- Week 24 | 6.1 [5.1 to 7.3] | 6.15 [5.03 to 7.43] | 6.05 [5 to 7.43] | 6.1 [5.01 to 7.43]
  WBC (1000 cells/cubic mm)- Week 32: number analyzed (Participants) | 802 | 797 | 788 | 1585
  WBC (1000 cells/cubic mm)- Week 32 | 6.1 [4.96 to 7.33] | 6.1 [5 to 7.4] | 6.05 [5 to 7.4] | 6.1 [5 to 7.4]
  WBC (1000 cells/cubic mm)- Week 40: number analyzed (Participants) | 790 | 786 | 765 | 1551
  WBC (1000 cells/cubic mm)- Week 40 | 6.09 [5 to 7.3] | 6.09 [4.9 to 7.3] | 5.95 [5 to 7.21] | 6 [4.9 to 7.25]
  WBC (1000 cells/cubic mm)- Week 48: number analyzed (Participants) | 772 | 775 | 753 | 1528
  WBC (1000 cells/cubic mm)- Week 48 | 6.16 [5.1 to 7.41] | 6 [5 to 7.21] | 6 [5.03 to 7.14] | 6 [5 to 7.18]
  WBC (1000 cells/cubic mm)- Week 56: number analyzed (Participants) | 754 | 763 | 750 | 1513
  WBC (1000 cells/cubic mm)- Week 56 | 6.1 [5.05 to 7.3] | 6.04 [4.88 to 7.43] | 5.9 [4.94 to 7.12] | 6 [4.9 to 7.3]
  WBC (1000 cells/cubic mm)- Week 64: number analyzed (Participants) | 737 | 748 | 721 | 1469
  WBC (1000 cells/cubic mm)- Week 64 | 6.05 [5.04 to 7.2] | 5.9 [4.9 to 7.38] | 5.95 [4.9 to 7.11] | 5.94 [4.9 to 7.2]
  WBC (1000 cells/cubic mm)- Week 72: number analyzed (Participants) | 722 | 731 | 719 | 1450
  WBC (1000 cells/cubic mm)- Week 72 | 5.91 [5 to 7.1] | 5.92 [4.89 to 7.2] | 6.05 [5 to 7.3] | 6 [4.9 to 7.22]
  Platelets (1000 cells/cubic mm)- Week 0: number analyzed (Participants) | 902 | 898 | 897 | 1795
  Platelets (1000 cells/cubic mm)- Week 0 | 248.5 [213 to 286] | 248 [210 to 289] | 249 [214 to 290] | 248.1 [212 to 290]
  Platelets (1000 cells/cubic mm)- Week 8: number analyzed (Participants) | 864 | 853 | 854 | 1707
  Platelets (1000 cells/cubic mm)- Week 8 | 248 [214.95 to 289] | 250 [213 to 291] | 248 [213 to 288] | 249 [213 to 290]
  Platelets (1000 cells/cubic mm)- Week 16: number analyzed (Participants) | 840 | 834 | 831 | 1665
  Platelets (1000 cells/cubic mm)- Week 16 | 249.5 [216 to 287] | 252 [214 to 293] | 251 [214 to 291] | 251 [214 to 292]
  Platelets (1000 cells/cubic mm)- Week 24: number analyzed (Participants) | 812 | 817 | 805 | 1622
  Platelets (1000 cells/cubic mm)- Week 24 | 251.5 [217 to 290.95] | 250 [215 to 292] | 251 [214 to 287] | 250.5 [214 to 289]
  Platelets (1000 cells/cubic mm)- Week 32: number analyzed (Participants) | 802 | 796 | 788 | 1584
  Platelets (1000 cells/cubic mm)- Week 32 | 252 [218 to 290] | 253.5 [216 to 296] | 250 [215 to 289] | 252 [215.75 to 291]
  Platelets (1000 cells/cubic mm)- Week 40: number analyzed (Participants) | 790 | 786 | 765 | 1551
  Platelets (1000 cells/cubic mm)- Week 40 | 250.7 [218 to 289] | 254.5 [215.3 to 294] | 250 [213 to 288] | 252 [214 to 291]
  Platelets (1000 cells/cubic mm)- Week 48: number analyzed (Participants) | 771 | 775 | 753 | 1528
  Platelets (1000 cells/cubic mm)- Week 48 | 251 [220 to 290] | 256 [219 to 291] | 251 [215 to 289] | 253 [217 to 290.2]
  Platelets (1000 cells/cubic mm)- Week 56: number analyzed (Participants) | 753 | 763 | 750 | 1513
  Platelets (1000 cells/cubic mm)- Week 56 | 254 [220 to 294] | 256 [219 to 296] | 251 [215 to 292] | 253 [217 to 294]
  Platelets (1000 cells/cubic mm)- Week 64: number analyzed (Participants) | 737 | 747 | 721 | 1468
  Platelets (1000 cells/cubic mm)- Week 64 | 254 [219 to 291] | 256 [219 to 296] | 249 [216 to 289] | 252 [217 to 293]
  Platelets (1000 cells/cubic mm)- Week 72: number analyzed (Participants) | 721 | 731 | 719 | 1450
  Platelets (1000 cells/cubic mm)- Week 72 | 254 [221 to 297] | 253 [220 to 298] | 253 [219 to 289] | 253 [219 to 293]

9. Primary Outcome: Chemistry and Hematology Laboratory Measures Meeting Grade 3 AE Criteria or Above
Description: The number (percentage) of participants with chemistry and hematology laboratory measures meeting grade 3 AE criteria or above as specified in the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017] is tabulated by treatment group and timepoint. Excludes measures taken prior to exposure to study product at Week 0/Infusion 1.
Time Frame: Measured at Weeks 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
Participants
  ALT (SGPT) (U/L)- Week 8: number analyzed (Participants) | 865 | 855 | 856 | 1711
  ALT (SGPT) (U/L)- Week 8 | 1 | 0 | 1 | 1
  ALT (SGPT) (U/L)- Week 16: number analyzed (Participants) | 841 | 836 | 832 | 1668
  ALT (SGPT) (U/L)- Week 16 | 1 | 0 | 4 | 4
  ALT (SGPT) (U/L)- Week 24: number analyzed (Participants) | 811 | 820 | 805 | 1625
  ALT (SGPT) (U/L)- Week 24 | 3 | 2 | 2 | 4
  ALT (SGPT) (U/L)- Week 32: number analyzed (Participants) | 802 | 797 | 787 | 1584
  ALT (SGPT) (U/L)- Week 32 | 2 | 1 | 1 | 2
  ALT (SGPT) (U/L)- Week 40: number analyzed (Participants) | 790 | 784 | 765 | 1549
  ALT (SGPT) (U/L)- Week 40 | 0 | 2 | 1 | 3
  ALT (SGPT) (U/L)- Week 48: number analyzed (Participants) | 772 | 776 | 754 | 1530
  ALT (SGPT) (U/L)- Week 48 | 4 | 0 | 1 | 1
  ALT (SGPT) (U/L)- Week 56: number analyzed (Participants) | 754 | 763 | 749 | 1512
  ALT (SGPT) (U/L)- Week 56 | 1 | 4 | 3 | 7
  ALT (SGPT) (U/L)- Week 64: number analyzed (Participants) | 737 | 748 | 722 | 1470
  ALT (SGPT) (U/L)- Week 64 | 3 | 2 | 1 | 3
  ALT (SGPT) (U/L)- Week 72: number analyzed (Participants) | 721 | 731 | 718 | 1449
  ALT (SGPT) (U/L)- Week 72 | 1 | 3 | 0 | 3
  Hemoglobin (g/dL)- Week 8: number analyzed (Participants) | 865 | 853 | 855 | 1708
  Hemoglobin (g/dL)- Week 8 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 16: number analyzed (Participants) | 841 | 836 | 832 | 1668
  Hemoglobin (g/dL)- Week 16 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 24: number analyzed (Participants) | 812 | 819 | 805 | 1624
  Hemoglobin (g/dL)- Week 24 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 32: number analyzed (Participants) | 802 | 797 | 788 | 1585
  Hemoglobin (g/dL)- Week 32 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 40: number analyzed (Participants) | 790 | 786 | 765 | 1551
  Hemoglobin (g/dL)- Week 40 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 48: number analyzed (Participants) | 772 | 775 | 753 | 1528
  Hemoglobin (g/dL)- Week 48 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 56: number analyzed (Participants) | 754 | 763 | 750 | 1513
  Hemoglobin (g/dL)- Week 56 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 64: number analyzed (Participants) | 737 | 748 | 721 | 1469
  Hemoglobin (g/dL)- Week 64 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 72: number analyzed (Participants) | 722 | 731 | 719 | 1450
  Hemoglobin (g/dL)- Week 72 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)- Week 8: number analyzed (Participants) | 866 | 855 | 856 | 1711
  Creatinine (mg/dL)- Week 8 | 7 | 1 | 2 | 3
  Creatinine (mg/dL)- Week 16: number analyzed (Participants) | 841 | 836 | 832 | 1668
  Creatinine (mg/dL)- Week 16 | 3 | 3 | 3 | 6
  Creatinine (mg/dL)- Week 24: number analyzed (Participants) | 812 | 820 | 805 | 1625
  Creatinine (mg/dL)- Week 24 | 6 | 3 | 2 | 5
  Creatinine (mg/dL)- Week 32: number analyzed (Participants) | 802 | 797 | 787 | 1584
  Creatinine (mg/dL)- Week 32 | 4 | 3 | 5 | 8
  Creatinine (mg/dL)- Week 40: number analyzed (Participants) | 791 | 786 | 765 | 1551
  Creatinine (mg/dL)- Week 40 | 5 | 7 | 6 | 13
  Creatinine (mg/dL)- Week 48: number analyzed (Participants) | 772 | 776 | 754 | 1530
  Creatinine (mg/dL)- Week 48 | 3 | 3 | 1 | 4
  Creatinine (mg/dL)- Week 56: number analyzed (Participants) | 754 | 763 | 750 | 1513
  Creatinine (mg/dL)- Week 56 | 5 | 4 | 2 | 6
  Creatinine (mg/dL)- Week 64: number analyzed (Participants) | 737 | 748 | 722 | 1470
  Creatinine (mg/dL)- Week 64 | 3 | 5 | 2 | 7
  Creatinine (mg/dL)- Week 72: number analyzed (Participants) | 722 | 732 | 718 | 1450
  Creatinine (mg/dL)- Week 72 | 4 | 4 | 2 | 6
  WBC (1000/cubic mm)- Week 8: number analyzed (Participants) | 865 | 853 | 855 | 1708
  WBC (1000/cubic mm)- Week 8 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Week 16: number analyzed (Participants) | 841 | 836 | 832 | 1668
  WBC (1000/cubic mm)- Week 16 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Week 24: number analyzed (Participants) | 812 | 819 | 805 | 1624
  WBC (1000/cubic mm)- Week 24 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Week 32: number analyzed (Participants) | 802 | 797 | 788 | 1585
  WBC (1000/cubic mm)- Week 32 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Week 40: number analyzed (Participants) | 790 | 786 | 765 | 1551
  WBC (1000/cubic mm)- Week 40 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Week 48: number analyzed (Participants) | 772 | 775 | 753 | 1528
  WBC (1000/cubic mm)- Week 48 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Week 56: number analyzed (Participants) | 754 | 763 | 750 | 1513
  WBC (1000/cubic mm)- Week 56 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Week 64: number analyzed (Participants) | 737 | 748 | 721 | 1469
  WBC (1000/cubic mm)- Week 64 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Week 72: number analyzed (Participants) | 722 | 731 | 719 | 1450
  WBC (1000/cubic mm)- Week 72 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 8: number analyzed (Participants) | 864 | 853 | 854 | 1707
  Platelets (1000/cubic mm)- Week 8 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 16: number analyzed (Participants) | 840 | 834 | 831 | 1665
  Platelets (1000/cubic mm)- Week 16 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 24: number analyzed (Participants) | 812 | 817 | 805 | 1622
  Platelets (1000/cubic mm)- Week 24 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 32: number analyzed (Participants) | 802 | 796 | 788 | 1584
  Platelets (1000/cubic mm)- Week 32 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 40: number analyzed (Participants) | 790 | 786 | 765 | 1551
  Platelets (1000/cubic mm)- Week 40 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 48: number analyzed (Participants) | 771 | 775 | 753 | 1528
  Platelets (1000/cubic mm)- Week 48 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 56: number analyzed (Participants) | 753 | 763 | 750 | 1513
  Platelets (1000/cubic mm)- Week 56 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 64: number analyzed (Participants) | 737 | 747 | 721 | 1468
  Platelets (1000/cubic mm)- Week 64 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Week 72: number analyzed (Participants) | 721 | 731 | 719 | 1450
  Platelets (1000/cubic mm)- Week 72 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 8: number analyzed (Participants) | 865 | 851 | 854 | 1705
  Lymphocytes (cells/cubic mm)- Week 8 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 16: number analyzed (Participants) | 840 | 836 | 832 | 1668
  Lymphocytes (cells/cubic mm)- Week 16 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 24: number analyzed (Participants) | 811 | 819 | 805 | 1624
  Lymphocytes (cells/cubic mm)- Week 24 | 1 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 32: number analyzed (Participants) | 802 | 797 | 788 | 1585
  Lymphocytes (cells/cubic mm)- Week 32 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 40: number analyzed (Participants) | 789 | 786 | 765 | 1551
  Lymphocytes (cells/cubic mm)- Week 40 | 0 | 0 | 1 | 1
  Lymphocytes (cells/cubic mm)- Week 48: number analyzed (Participants) | 772 | 774 | 752 | 1526
  Lymphocytes (cells/cubic mm)- Week 48 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 56: number analyzed (Participants) | 754 | 762 | 750 | 1512
  Lymphocytes (cells/cubic mm)- Week 56 | 1 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 64: number analyzed (Participants) | 737 | 748 | 721 | 1469
  Lymphocytes (cells/cubic mm)- Week 64 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 72: number analyzed (Participants) | 722 | 731 | 719 | 1450
  Lymphocytes (cells/cubic mm)- Week 72 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 8: number analyzed (Participants) | 865 | 851 | 854 | 1705
  Neutrophils (cells/cubic mm)- Week 8 | 0 | 1 | 0 | 1
  Neutrophils (cells/cubic mm)- Week 16: number analyzed (Participants) | 840 | 836 | 832 | 1668
  Neutrophils (cells/cubic mm)- Week 16 | 0 | 1 | 0 | 1
  Neutrophils (cells/cubic mm)- Week 24: number analyzed (Participants) | 811 | 819 | 805 | 1624
  Neutrophils (cells/cubic mm)- Week 24 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 32: number analyzed (Participants) | 802 | 797 | 788 | 1585
  Neutrophils (cells/cubic mm)- Week 32 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 40: number analyzed (Participants) | 789 | 786 | 765 | 1551
  Neutrophils (cells/cubic mm)- Week 40 | 0 | 1 | 0 | 1
  Neutrophils (cells/cubic mm)- Week 48: number analyzed (Participants) | 772 | 774 | 752 | 1526
  Neutrophils (cells/cubic mm)- Week 48 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 56: number analyzed (Participants) | 754 | 762 | 750 | 1512
  Neutrophils (cells/cubic mm)- Week 56 | 0 | 1 | 0 | 1
  Neutrophils (cells/cubic mm)- Week 64: number analyzed (Participants) | 737 | 748 | 721 | 1469
  Neutrophils (cells/cubic mm)- Week 64 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 72: number analyzed (Participants) | 722 | 731 | 719 | 1450
  Neutrophils (cells/cubic mm)- Week 72 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Early Infusion Discontinuation and Reasons for Discontinuation
Description: The number (percentage) of participants with early permanent discontinuation of infusions and their reason for discontinuation is summarized by treatment group. Includes all discontinuations documented on a study case report form.
Time Frame: Measured through Week 72 (the last infusion visit).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 903 | 899 | 897 | 1796
Participants
  Pregnancy | 0 | 0 | 0 | 0
  HIV infection | 37 | 32 | 21 | 53
  Death | 0 | 2 | 0 | 2
  Clinical event other than reactogenicity | 14 | 16 | 20 | 36
  Reactogenicity Symptom | 0 | 0 | 0 | 0
  Investigator Reason | 7 | 2 | 1 | 3
  Participant refused study product infusion | 5 | 5 | 7 | 12
  Co-enrollment in a study | 1 | 2 | 1 | 3
  Two(2) reactive HIV tests | 0 | 0 | 3 | 3
  Other | 11 | 6 | 7 | 13
  Termination from study for non-medical reason(s) | 69 | 75 | 80 | 155
  No Discontinuation | 759 | 759 | 757 | 1516

11. Primary Outcome: Incidence Rate of Early Infusion Discontinuation
Description: Incidence rate (95% CI) of early infusion discontinuation per 100 person years. Includes discontinuations documented on a study case report form and operational discontinuations defined as 20 consecutive weeks without participant contact. Discontinuations due to pregnancy, death, or HIV-1 infection are right-censored.
Time Frame: Measured through Week 72 (the last infusion visit).
Population: Safety population
Measure: Number (95% Confidence Interval); unit: events per 100 person years
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01
Number analyzed (Participants) | 903 | 899 | 897
events per 100 person years | 8.9 [7.3 to 10.7] | 10 [8.3 to 11.9] | 8.8 [7.2 to 10.6]

12. Primary Outcome: Number of Participants With Documented HIV-1 Infection by the Week 80 Visit
Description: Prevention efficacy (PE) is measured as 1 minus the ratio (VRC01:control) of cumulative incidences of HIV-1 infection diagnosis between enrollment and the week 80 visit for assessment of the primary efficacy end point. Cumulative incidence was estimated with the Nelson-Aalen estimator for the cumulative hazard function, with stratification according to VRC01 dose and trial.
Time Frame: Measured through Week 80.
Population: MITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 898 | 895 | 894 | 1789
Participants | 38 | 32 | 28 | 60
Statistical Analysis 1: Comparison: Placebo vs Pooled VRC01; The primary PE analysis tests the null hypothesis PE equal to zero versus the alternative hypothesis PE not equal to zero using a 2-sided alpha equal 0.05 level Wald test of the equality of log cumulative hazard functions at the week 80 visit for the pooled VRC01 group versus the placebo group; Test type: Other; p = 0.15, wald — The threshold for statistical significance was p = 0.05; Prevention Efficacy (PE) = 26.6, 95% CI 2-sided [-11.7 to 51.8]
Statistical Analysis 2: Comparison: Placebo vs Low-Dose VRC01; A secondary analysis assesses the overall PE of the low-dose VRC01 group versus the placebo group; Test type: Other; Prevention Efficacy (PE) = 22.4, 95% CI 2-sided [-25.5 to 52.0]
Statistical Analysis 3: Comparison: Placebo vs High-Dose VRC01; A secondary analysis assesses the overall PE of the high-dose VRC01 group versus the placebo group; Test type: Other; Prevention Efficacy (PE) = 30.9, 95% CI 2-sided [-13.9 to 58.0]

13. Secondary Outcome: Serum Concentration of VRC01 in Participants Assigned to Receive the mAb
Description: The pharmacokinetic analyses of VRC01 involved a subgroup of VRC01 recipients who had not acquired HIV-1 infection through the week 88 visit and were not likely to have used preexposure prophylaxis (on the basis of self-report or testing of dried blood-spot samples), randomly sampled among the trials and dose groups. Midpoint and trough concentrations are the participant-level median concentrations at the 4-week and 8-week postinfusion visits, respectively, across all 10 infusion intervals.
Time Frame: Day 61 (5 days post infusion #2), Midpoint (4-weeks post infusion visits): Weeks 4, 12, 16, 28, 36, 44, 52, 60, 68, 76 and Trough (infusion visits): Pre dose at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
Population: Pilot study population
Measure: Median (Full Range); unit: μg/ml
Arm/Group | Low-Dose VRC01 | High-Dose VRC01
Number analyzed (Participants) | 12 | 12
μg/ml
  4-week post infusion visit | 23.1 [8.8 to 43.9] | 55.1 [26.6 to 89.5]
  8-week post infusion visit | 5.8 [1.5 to 18.3] | 15.4 [4.5 to 29.8]
  Day 61 | 65.7 [41.7 to 116.1] | 212 [125.5 to 287.5]

14. Secondary Outcome: VRC01 Clinical Lot Neutralization of Founder Viruses (IC80)
Description: The VRC01 80% inhibitory concentration (IC80) of acquired isolates was measured with the TZM-bl assay using the earliest available post-HIV-infection serum sample. Median and IQR are summarized immediately below, then the analysis of prevention efficacy was repeated for each of three prespecified categories of in vitro susceptibility of the infecting strain (IC80 less than 1 μg per milliliter, 1 to 3 μg per milliliter, or >3 μg per milliliter) with the use of the Aalen-Johansen estimator.
Time Frame: Measured through Week 80.
Population: MITT population
Measure: Median (Inter-Quartile Range); unit: μg/ml
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 898 | 895 | 894 | 1789
μg/ml | 3.28 [0.79 to 8.58] | 4.7 [2.39 to 19.43] | 5.78 [2.3 to 12.56] | 4.97 [2.34 to 15.86]
Statistical Analysis 1: Comparison: Placebo vs Pooled VRC01; PE against IC80 of least sensitive variant less than 1; Test type: Other; Prevention Efficacy (PE) = 73, 95% CI 2-sided [27.6 to 89.9]
Statistical Analysis 2: Comparison: Placebo vs Pooled VRC01; PE against IC80 of least sensitive variant 1-3; Test type: Other; Prevention Efficacy (PE) = 6.1, 95% CI 2-sided [-174.3 to 67.8]
Statistical Analysis 3: Comparison: Placebo vs Pooled VRC01; PE against IC80 of least sensitive variant > 3; Test type: Other; Prevention Efficacy (PE) = 8.6, 95% CI 2-sided [-68.1 to 50.3]

15. Secondary Outcome: VRC01 Serum Neutralization of Autologous Founder Viruses (ID50, ID80)
Description: Autologous titer (ID50, ID80) summaries, based on most sensitive virus, for first RNA+ samples from a subset of HIV-infected VRC01 recipients. Values below the limit of detection (less than 10) were set to NA. Summaries are only computed for the Pooled VRC01 arm.
Time Frame: First RNA+ Sample detected from baseline up to Week 104.
Population: Subset of HIV-infected VRC01 recipients
Measure: Median (Full Range); unit: titer
Arm/Group | Pooled VRC01
Number analyzed (Participants) | 31
titer
  ID50 | NA [NA to 125.3] — Values below the limit of detection (less than 10) were set to NA.
  ID80 | NA [NA to 34.18] — Values below the limit of detection (less than 10) were set to NA.

ADVERSE EVENTS:
Time Frame: The AE reporting period for this study comprises the entire study period for each individual participant (from study enrollment until study completion at the week 104 visit or discontinuation of the study)
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
All-Cause Mortality (participants affected / at risk) | 2/903 | 3/899 | 0/897 | 3/1796
Serious Adverse Events (participants affected / at risk) | 32/903 | 35/899 | 32/897 | 67/1796
Other Adverse Events (participants affected / at risk) | 750/903 | 771/899 | 742/897 | 1513/1796
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=903) | Low-Dose VRC01 (N=899) | High-Dose VRC01 (N=897) | Pooled VRC01 (N=1796)
Any Event in SOC (Cardiac disorders) | 1 (1) | 0 (0) | 3 (4) | 3 (4)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Gastrointestinal disorders) | 3 (6) | 0 (0) | 4 (5) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Infections and infestations) | 10 (10) | 14 (15) | 10 (10) | 24 (25)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 4 (4) | 5 (5) | 3 (3) | 8 (8)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 5 (8) | 7 (8) | 2 (2) | 9 (10)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Psychiatric disorders) | 10 (18) | 8 (10) | 12 (15) | 20 (25)
Alcoholism (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 2 (3) | 3 (4) | 5 (7)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Emotional distress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Substance dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4) | 5 (5)
Suicide attempt (Psychiatric disorders) | 4 (6) | 2 (2) | 2 (2) | 4 (4)
Any Event in SOC (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=903) | Low-Dose VRC01 (N=899) | High-Dose VRC01 (N=897) | Pooled VRC01 (N=1796)
Any Event in SOC (Blood and lymphatic system disorders) | 17 (18) | 26 (28) | 23 (29) | 49 (57)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 11 (12) | 15 (16) | 14 (17) | 29 (33)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Microcytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 5 (6) | 8 (9)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Cardiac disorders) | 7 (8) | 3 (3) | 3 (3) | 6 (6)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brugada syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intracardiac mass (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Congenital, familial and genetic disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Encephalocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Frenulum breve (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tourette's disorder (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 12 (12) | 17 (19) | 5 (5) | 22 (24)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 7 (7) | 1 (1) | 8 (8)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 2 (2) | 1 (1) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Eye disorders) | 14 (14) | 11 (12) | 8 (8) | 19 (20)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Eye pain (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Keratoconus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lagophthalmos (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Scintillating scotoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Gastrointestinal disorders) | 155 (211) | 183 (269) | 175 (253) | 358 (522)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1) | 7 (7) | 8 (8)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 8 (8) | 11 (11) | 19 (19)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 5 (5) | 4 (4) | 9 (9)
Acquired oesophageal web (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 4 (5) | 10 (12) | 8 (8) | 18 (20)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 8 (8) | 3 (4) | 3 (3) | 6 (7)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Anorectal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
Aphthous ulcer (Gastrointestinal disorders) | 5 (5) | 5 (5) | 2 (2) | 7 (7)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (5) | 5 (6) | 9 (11)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (2) | 4 (4) | 6 (7) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 57 (64) | 49 (62) | 58 (66) | 107 (128)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 3 (3) | 9 (9) | 12 (12)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Food poisoning (Gastrointestinal disorders) | 12 (12) | 18 (18) | 15 (16) | 33 (34)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 5 (5) | 5 (6) | 4 (4) | 9 (10)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (9) | 5 (5) | 10 (10) | 15 (15)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 11 (11) | 21 (23) | 10 (10) | 31 (33)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertrophy of tongue papillae (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip erosion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malpositioned teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Mouth cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 10 (10) | 18 (19) | 16 (18) | 34 (37)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
Oral papule (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Proctitis (Gastrointestinal disorders) | 5 (6) | 8 (11) | 8 (9) | 16 (20)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 6 (6) | 2 (2) | 8 (8)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Tooth demineralisation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 5 (5)
Toothache (Gastrointestinal disorders) | 6 (6) | 8 (9) | 10 (10) | 18 (19)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (7) | 4 (4) | 11 (11)
Any Event in SOC (General disorders) | 65 (77) | 88 (106) | 80 (93) | 168 (199)
Adverse drug reaction (General disorders) | 4 (4) | 4 (4) | 7 (7) | 11 (11)
Adverse food reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Axillary pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Chills (General disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 11 (11) | 13 (13) | 12 (13) | 25 (26)
Feeling hot (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hangover (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 37 (38) | 36 (39) | 36 (39) | 72 (78)
Infusion site bruising (General disorders) | 0 (0) | 3 (5) | 1 (1) | 4 (6)
Infusion site extravasation (General disorders) | 3 (3) | 7 (7) | 2 (2) | 9 (9)
Infusion site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lithiasis (General disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Malaise (General disorders) | 0 (0) | 4 (4) | 1 (1) | 5 (5)
Nodule (General disorders) | 0 (0) | 3 (3) | 3 (3) | 6 (6)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3) | 3 (3) | 6 (6)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 4 (4) | 2 (2) | 6 (6)
Peripheral swelling (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 8 (8) | 4 (4) | 12 (12)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Hepatobiliary disorders) | 5 (5) | 7 (8) | 2 (3) | 9 (11)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deficiency of bile secretion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Hepatitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Immune system disorders) | 23 (25) | 19 (20) | 12 (13) | 31 (33)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 4 (5) | 0 (0) | 3 (3) | 3 (3)
Food allergy (Immune system disorders) | 4 (5) | 3 (3) | 1 (1) | 4 (4)
Hypersensitivity (Immune system disorders) | 3 (3) | 5 (5) | 1 (1) | 6 (6)
Jarisch-Herxheimer reaction (Immune system disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Mite allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 10 (10) | 9 (9) | 6 (6) | 15 (15)
Any Event in SOC (Infections and infestations) | 591 (1612) | 612 (1732) | 585 (1669) | 1197 (3401)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 6 (6) | 5 (5) | 6 (6) | 11 (11)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acariasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 19 (20) | 18 (21) | 17 (19) | 35 (40)
Acute hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Amoebic dysentery (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Anal chlamydia infection (Infections and infestations) | 162 (211) | 176 (244) | 187 (244) | 363 (488)
Anal fistula infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fungal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal human papilloma virus infection (Infections and infestations) | 1 (2) | 2 (2) | 4 (4) | 6 (6)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascariasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Balanitis candida (Infections and infestations) | 3 (6) | 2 (2) | 1 (1) | 3 (3)
Blastocystis infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 8 (9) | 3 (3) | 7 (7) | 10 (10)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 12 (13) | 14 (14) | 12 (13) | 26 (27)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Burn infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 7 (9) | 3 (3) | 6 (6) | 9 (9)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cestode infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chancroid (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chlamydial infection (Infections and infestations) | 9 (12) | 4 (4) | 10 (12) | 14 (16)
Cholera (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 6 (6) | 11 (11) | 11 (11) | 22 (22)
Conjunctivitis bacterial (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 3 (3)
Conjunctivitis viral (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatophytosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 5 (5) | 2 (2) | 4 (4) | 6 (6)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysentery (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 3 (3) | 3 (3) | 4 (6) | 7 (9)
Ear infection bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Erythema migrans (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 5 (5) | 4 (4) | 3 (3) | 7 (7)
Folliculitis (Infections and infestations) | 12 (12) | 10 (10) | 9 (9) | 19 (19)
Fungal balanitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 4 (4)
Fungal skin infection (Infections and infestations) | 2 (2) | 4 (4) | 5 (5) | 9 (9)
Furuncle (Infections and infestations) | 2 (2) | 1 (1) | 4 (5) | 5 (6)
Gastroenteritis (Infections and infestations) | 48 (53) | 43 (49) | 38 (44) | 81 (93)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 12 (12) | 4 (4) | 16 (16)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 7 (8) | 7 (9) | 11 (14) | 18 (23)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 2 (3)
Genital candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Genital herpes (Infections and infestations) | 8 (8) | 13 (16) | 10 (10) | 23 (26)
Genital herpes simplex (Infections and infestations) | 5 (5) | 4 (4) | 4 (4) | 8 (8)
Genitourinary chlamydia infection (Infections and infestations) | 50 (54) | 46 (54) | 43 (46) | 89 (100)
Genitourinary tract gonococcal infection (Infections and infestations) | 35 (37) | 35 (42) | 36 (37) | 71 (79)
Giardiasis (Infections and infestations) | 3 (3) | 3 (4) | 4 (4) | 7 (8)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Gingivitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 4 (4)
Gonococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gonorrhoea (Infections and infestations) | 6 (6) | 4 (4) | 7 (7) | 11 (11)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 6 (6) | 0 (0) | 6 (6)
Hepatitis C (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 4 (4) | 9 (11) | 13 (15)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 3 (5) | 1 (1) | 4 (6)
Hordeolum (Infections and infestations) | 7 (7) | 8 (14) | 6 (6) | 14 (20)
Impetigo (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 5 (5)
Infected bite (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Infection parasitic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Infective corneal ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 17 (17) | 16 (17) | 11 (12) | 27 (29)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 3 (4) | 1 (1) | 4 (5) | 5 (6)
Latent syphilis (Infections and infestations) | 20 (21) | 25 (28) | 19 (20) | 44 (48)
Latent tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lice infestation (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 5 (5)
Localised infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphadenitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphogranuloma venereum (Infections and infestations) | 1 (1) | 3 (3) | 5 (5) | 8 (8)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Nasopharyngitis (Infections and infestations) | 53 (65) | 55 (75) | 51 (72) | 106 (147)
Neurosyphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nipple infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 3 (3) | 6 (6) | 3 (3) | 9 (9)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 10 (11) | 8 (8) | 6 (6) | 14 (14)
Oral pustule (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal gonococcal infection (Infections and infestations) | 51 (61) | 65 (77) | 69 (79) | 134 (156)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 6 (6)
Otitis media acute (Infections and infestations) | 0 (0) | 3 (3) | 4 (4) | 7 (7)
Papilloma viral infection (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 2 (2)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Paronychia (Infections and infestations) | 2 (3) | 3 (3) | 0 (0) | 3 (3)
Parotitis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Penile abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pericoronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal chlamydia infection (Infections and infestations) | 11 (11) | 12 (14) | 6 (8) | 18 (22)
Pharyngitis (Infections and infestations) | 31 (34) | 25 (26) | 26 (31) | 51 (57)
Pharyngitis bacterial (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 5 (5)
Pharyngitis streptococcal (Infections and infestations) | 30 (34) | 25 (28) | 26 (31) | 51 (59)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 5 (5)
Pilonidal cyst (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Primary syphilis (Infections and infestations) | 6 (6) | 10 (10) | 5 (5) | 15 (15)
Proctitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Proctitis gonococcal (Infections and infestations) | 124 (152) | 121 (151) | 125 (146) | 246 (297)
Proctitis herpes (Infections and infestations) | 5 (5) | 4 (4) | 2 (3) | 6 (7)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Puncture site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pustule (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 5 (5) | 8 (8)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 5 (5)
Schistosomiasis cutaneous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secondary syphilis (Infections and infestations) | 4 (4) | 8 (8) | 7 (7) | 15 (15)
Sexually transmitted disease (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 33 (37) | 31 (38) | 31 (36) | 62 (74)
Sinusitis bacterial (Infections and infestations) | 2 (2) | 3 (3) | 1 (2) | 4 (5)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 3 (3) | 2 (3) | 4 (4) | 6 (7)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Strongyloidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Syphilis (Infections and infestations) | 52 (55) | 74 (79) | 76 (78) | 150 (157)
Syphilis anal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syphilis genital (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 6 (6) | 3 (4) | 7 (7) | 10 (11)
Tinea faciei (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 4 (5) | 2 (2) | 6 (7)
Tinea pedis (Infections and infestations) | 2 (2) | 7 (7) | 4 (4) | 11 (11)
Tinea versicolour (Infections and infestations) | 4 (5) | 1 (1) | 4 (5) | 5 (6)
Tonsillitis (Infections and infestations) | 11 (12) | 15 (15) | 15 (17) | 30 (32)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 3 (3) | 1 (1) | 10 (10) | 11 (11)
Tooth infection (Infections and infestations) | 11 (12) | 11 (11) | 7 (8) | 18 (19)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 185 (285) | 160 (248) | 182 (280) | 342 (528)
Upper respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 4 (4)
Urethral discharge syndrome (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Urethritis (Infections and infestations) | 13 (17) | 22 (25) | 30 (31) | 52 (56)
Urethritis chlamydial (Infections and infestations) | 13 (13) | 21 (21) | 10 (10) | 31 (31)
Urethritis gonococcal (Infections and infestations) | 13 (13) | 12 (13) | 9 (9) | 21 (22)
Urethritis mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 11 (11) | 11 (11) | 10 (11) | 21 (22)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vaginitis chlamydial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 27 (35) | 38 (44) | 32 (36) | 70 (80)
Viral pharyngitis (Infections and infestations) | 8 (11) | 7 (9) | 3 (3) | 10 (12)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Viral tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 22 (26) | 34 (46) | 29 (35) | 63 (81)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginitis gonococcal (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Wound infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 117 (160) | 138 (194) | 127 (172) | 265 (366)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Animal bite (Injury, poisoning and procedural complications) | 4 (4) | 8 (8) | 1 (1) | 9 (9)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 14 (15) | 4 (4) | 10 (10) | 14 (14)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Barotitis media (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Breast injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Burn oral cavity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Burns second degree (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chemical burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 3 (4) | 4 (4) | 4 (4) | 8 (8)
Contusion (Injury, poisoning and procedural complications) | 13 (13) | 15 (17) | 11 (11) | 26 (28)
Corneal abrasion (Injury, poisoning and procedural complications) | 2 (2) | 3 (4) | 0 (0) | 3 (4)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 2 (3) | 1 (2) | 0 (0) | 1 (2)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (6) | 6 (6) | 11 (12)
Genital contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (3) | 6 (6)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 0 (0) | 3 (3)
Human bite (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 1 (1) | 3 (4)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 4 (4) | 6 (6)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 2 (2) | 6 (6)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 14 (16) | 18 (19) | 7 (7) | 25 (26)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 3 (3) | 6 (6)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Mallet finger (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 6 (6) | 18 (19) | 16 (16) | 34 (35)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Penis injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (2) | 2 (3)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 5 (6) | 8 (9) | 18 (23) | 26 (32)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 9 (9) | 15 (17) | 4 (4) | 19 (21)
Skin laceration (Injury, poisoning and procedural complications) | 11 (12) | 20 (22) | 10 (10) | 30 (32)
Skin scar contracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 5 (6) | 4 (4) | 8 (8) | 12 (12)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 6 (6) | 8 (8)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urethral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Venomous sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 4 (4) | 6 (6)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Any Event in SOC (Investigations) | 323 (659) | 331 (618) | 319 (575) | 650 (1193)
Alanine aminotransferase increased (Investigations) | 193 (321) | 187 (282) | 172 (265) | 359 (547)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 26 (37) | 21 (29) | 22 (28) | 43 (57)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 2 (3) | 3 (4) | 5 (7)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 6 (8) | 7 (12) | 5 (5) | 12 (17)
Blood cholesterol increased (Investigations) | 3 (5) | 0 (0) | 2 (2) | 2 (2)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 106 (146) | 101 (141) | 117 (152) | 218 (293)
Blood glucose decreased (Investigations) | 1 (1) | 2 (3) | 1 (1) | 3 (4)
Blood glucose increased (Investigations) | 7 (13) | 11 (14) | 12 (16) | 23 (30)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 32 (51) | 34 (48) | 28 (46) | 62 (94)
Blood testosterone decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 3 (4) | 0 (0) | 2 (2) | 2 (2)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Creatinine renal clearance increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate abnormal (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 4 (4) | 8 (9) | 5 (6) | 13 (15)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymph node palpable (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (4) | 3 (3) | 7 (7)
Neutrophil count decreased (Investigations) | 16 (21) | 27 (43) | 14 (22) | 41 (65)
Platelet count decreased (Investigations) | 7 (11) | 8 (8) | 5 (6) | 13 (14)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 2 (2) | 3 (3) | 2 (2) | 5 (5)
Prothrombin time prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Red blood cell schistocytes present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 4 (4) | 5 (9) | 2 (4) | 7 (13)
Any Event in SOC (Metabolism and nutrition disorders) | 12 (12) | 20 (21) | 17 (21) | 37 (42)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Dairy intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 2 (2) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 2 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3) | 6 (6)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 3 (3) | 5 (5)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 97 (130) | 121 (160) | 95 (143) | 216 (303)
Ankle impingement (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (26) | 34 (36) | 30 (34) | 64 (70)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (34) | 27 (30) | 31 (36) | 58 (66)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 4 (5) | 7 (8)
Coccydynia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 0 (0) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 2 (2) | 8 (8)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 3 (3) | 8 (8)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (3) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 20 (24) | 11 (11) | 31 (35)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9) | 8 (8) | 17 (17)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (17) | 16 (17) | 21 (22) | 37 (39)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 0 (0) | 3 (3)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 3 (3) | 6 (6)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (20) | 18 (21) | 13 (14) | 31 (35)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 7 (8) | 8 (8) | 15 (16)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 1 (1) | 5 (5)
Any Event in SOC (Nervous system disorders) | 47 (56) | 65 (78) | 61 (76) | 126 (154)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
Circadian rhythm sleep disorder (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7) | 9 (9) | 5 (6) | 14 (15)
Headache (Nervous system disorders) | 22 (22) | 23 (25) | 27 (33) | 50 (58)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 3 (3) | 6 (9) | 1 (1) | 7 (10)
Nerve compression (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Nerve degeneration (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 5 (6) | 7 (8)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 5 (5) | 11 (11) | 5 (5) | 16 (16)
Sciatica (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 4 (4)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 1 (1) | 6 (6) | 7 (7)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Any Event in SOC (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 56 (78) | 56 (73) | 58 (75) | 114 (148)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Alcohol use disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 16 (16) | 13 (13) | 29 (29)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 2 (2) | 3 (3) | 2 (2) | 5 (5)
Bipolar II disorder (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Borderline personality disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bruxism (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 15 (15) | 19 (20) | 19 (19) | 38 (39)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug abuse (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Grief reaction (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 11 (11) | 5 (5) | 11 (12) | 16 (17)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Panic attack (Psychiatric disorders) | 3 (5) | 4 (4) | 3 (3) | 7 (7)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Seasonal affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Social anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Stress (Psychiatric disorders) | 0 (0) | 4 (4) | 5 (5) | 9 (9)
Substance abuse (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 5 (5) | 5 (5) | 4 (4) | 9 (9)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 87 (106) | 86 (117) | 91 (109) | 177 (226)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Costovertebral angle tenderness (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 16 (16) | 18 (19) | 12 (13) | 30 (32)
Glomerulonephritis chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 2 (2) | 5 (6) | 2 (2) | 7 (8)
Haematuria (Renal and urinary disorders) | 29 (32) | 34 (43) | 28 (36) | 62 (79)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 6 (7) | 9 (9) | 15 (16)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 29 (35) | 19 (23) | 28 (30) | 47 (53)
Renal colic (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sterile pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 8 (9) | 8 (8) | 11 (12) | 19 (20)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 40 (45) | 31 (33) | 37 (42) | 68 (75)
Balanoposthitis (Reproductive system and breast disorders) | 5 (5) | 5 (5) | 9 (9) | 14 (14)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Galactorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Genital discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital macule (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genital odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genital paraesthesia (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Genital ulceration (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nipple inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile blister (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Penile discharge (Reproductive system and breast disorders) | 9 (9) | 5 (6) | 7 (8) | 12 (14)
Penile erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Penile rash (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Penis disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 4 (4) | 3 (3) | 3 (3) | 6 (6)
Pruritus genital (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Scrotal dermatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (2) | 2 (2) | 2 (2) | 4 (4)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 76 (91) | 69 (87) | 80 (100) | 149 (187)
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3) | 5 (6) | 7 (9)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (11) | 15 (17) | 26 (28)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (2) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 7 (7) | 13 (13)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discolouration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 24 (28) | 29 (35) | 53 (63)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (5) | 2 (5) | 7 (10)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 5 (5) | 9 (10)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 6 (6) | 9 (9)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (4) | 6 (7)
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 100 (121) | 136 (165) | 118 (146) | 254 (311)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (11) | 3 (3) | 13 (14)
Acne cystic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 3 (3) | 5 (5)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 6 (6) | 10 (10)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 13 (14) | 20 (20) | 16 (17) | 36 (37)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 3 (3) | 8 (8)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 8 (8) | 11 (11)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Milia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (9) | 11 (14) | 19 (23)
Pemphigus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pityriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (4) | 5 (5) | 9 (9)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 11 (11) | 21 (22) | 7 (7) | 28 (29)
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (8) | 2 (2) | 10 (10)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 3 (3) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 4 (4)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (6) | 5 (6) | 9 (12)
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4) | 7 (7) | 11 (11)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 4 (4)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 3 (4)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 12 (13) | 16 (16) | 22 (26) | 38 (42)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Social circumstances) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Physical assault (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Victim of sexual abuse (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Vascular disorders) | 16 (17) | 9 (9) | 8 (9) | 17 (18)
Flushing (Vascular disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 13 (13) | 6 (6) | 3 (3) | 9 (9)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT02716675/Prot_001.pdf
  • Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT02716675/SAP_002.pdf
  • Informed Consent Form (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT02716675/ICF_000.pdf